CLINICAL TRIAL: NCT05810051
Title: Effects of a Cardiac Rehabilitation Program on Health-related Quality of Life in Patients With Coronary Microvascular Disease.
Brief Title: Exercise and Coronary Microvascular Disease
Acronym: ExerciseCMD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CoreAalst BV (Industry)
Collaborators: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA-021
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Coronary Microvascular Disease
Keywords: Exercise training
MeSH Terms: conditions — Microvascular Angina | interventions — Cardiac Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Optimal medical therapy (OMT) plus a program of cardiac rehabilitation (CR) (Experimental): The intervention group will receive cardiac rehabilitation in addition to lifestyle changes and pharmacological treatment.
  Interventions: Behavioral: Cardiac rehabilitation
- Optimal medical therapy (OMT) (No Intervention): The control group will be randomized to lifestyle changes and pharmacological treatment.
  In the 7 to 14 days after randomization optimal medical therapy will be started.

INTERVENTIONS:
Behavioral: Cardiac rehabilitation — The patients in this arm will be trained for 1 hour, 2 or 3 times per week for 36 sessions. In addition to the training program, the patients also get access to the cardiovascular educational program.
  The training (a 1h session) consists of 60% cardiovascular endurance training and 40% resistance training.
  Arms: Optimal medical therapy (OMT) plus a program of cardiac rehabilitation (CR)

SUMMARY:
Exercise CMD is a prospective single-center, open-label, parallel arms randomized controlled trial.

This trial aims to assess the impact of cardiac rehabilitation on top of optimal medical therapy on patient-reported outcomes in subjects with coronary microvascular disease and non-obstructive coronary artery disease.

Patients will undergo a microvascular assessment using bolus thermodilution techniques and those with criteria for microvascular angina (IMR ≥ 25) will be invited to participate.

Patients will be randomized in a 1:1 ratio to either optimal medical therapy (OMT) or OMT plus a program of cardiac rehabilitations (CR).

After randomization, spiro-ergometry and a SAQ-19 will be performed in all patients. Medical therapy will be standardized in both arms and the CR group will follow 36 sessions of the personalized physical training program of cardiac rehabilitation.

Approximately 204 subjects (102 in each group) will be included at one site (OLV Aalst, Belgium).

Clinical Follow-Up will be planned at 4 months. Patients with CCTA performed in standard of care will be invited for control CCTA 6 +/- 1 month after the invasive procedure.

ELIGIBILITY:
Inclusion Criteria:

* Non obstructive CAD (diameter stenosis <50% visual or FFR > 0.80)
* Angina at presentation
* Evidence of microvascular dysfunction (IMR ≥ 25)

Exclusion Criteria:

* Inability to give consent
* Acute coronary syndrome (ACS)
* Severe valve disease
* Permanent AF
* History of coronary artery bypass grafting (CABG)
* Cardiomyopathies
* Intolerance to adenosine
* Hemodynamic instability
* Not able to exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2023-07-31 (Actual); Primary Completion 2026-04-15 (Estimated); Study Completion 2027-10-15 (Estimated)

PRIMARY OUTCOMES:
Mean change in health-related Seattle Angina Questionnaire (SAQ19) between baseline and 4 months | 4 Months
  Mean change in health-related quality of life questionnaire as assessed by the Seattle Angina Questionnaire 19, between baseline and 4 months (SAQ-19 Summary Score) with a maximum score of 100 representing a good quality of life.

SECONDARY OUTCOMES:
Mean change in Seattle Angina Questionnaire (SAQ19)frequency score between baseline and 4 months | 4 Months
  Mean change in the Seattle Angina Questionnaire frequency score between baseline and 4 months with a maximum score of 100 representing no angina symptoms.
Mean change in VO2 peak between baseline and 4 months | 4 Months
  Mean change in exercise capacity, as assessed by the peak oxygen consumption (VO2 peak) derived from spiro-ergometry test between baseline and 4 months
Mean change in VE/VCO2 slope between baseline and 4 months | 4 Months
  Mean change in ventilatory efficiency, as assessed by the VE/VCO2 slope derived from spiro-ergometry test, between baseline and 4 months
Mean change in METS between baseline and 4 months | 4 Months
  Mean change in Metabole equivalents (METS) derived from spiro-ergometry test between baseline and 4 months
Mean change in health related quality of life assessed by the EuroQoL 5 dimensions - 5 levels (EQ5D-5L) Questionnaire between baseline and 4 months | 4 Months
  Mean change in health related quality of life as assessed by the EuroQoL 5 dimensions - 5 levels EQ5D-5L Index score between baseline and 4 months with a score of 1 representing a perfect health condition.
Mean change in vessel volume between patients randomized to exercise and controls | 6 Months
  Mean change in vessel volume as assessed by coronary CT angiography between patients randomized to exercise and controls (only for patients with baseline coronary CT angiography).

CONTACTS AND LOCATIONS:
Locations (1):
- OLV Aalst, Aalst, East-Flanders, Belgium